CLINICAL TRIAL: NCT05626023
Title: A Phase I Study to Evaluate the Safety and Tolerability of Human TH-SC01 Cell Injection for the Treatment of Perianal Fistulas in Crohn's Disease
Brief Title: A Study of Human TH-SC01 Cell Injection for Treating Perianal Fistulas in Patients With Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TH-SC 2.0
Record Dates: First submitted 2022-10-26; First posted 2022-11-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Perianal Fistula; Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human TH-SC01 cell injection (Experimental): Single injection of 0.6×10^7, 1.2×10^8, 1.8×10^8 cells/kg
  Interventions: Drug: Human TH-SC01 cell injection

INTERVENTIONS:
Drug: Human TH-SC01 cell injection — Single injection of human TH-SC01 cell injection

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of human TH-SC01 cell injection for the treatment of perianal fistulas in Crohn's Disease

DETAILED DESCRIPTION:
This study is a phase 1, single-arm, safety and tolerability study of human TH-SC01 cell injection for perianal fistulas in Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Subjects with Crohn's disease diagnosed at least 6 months earlier according to the Chinese Consensus Opinion on the Diagnosis and Treatment of Inflammatory Bowel Diseases (Beijing, 2018).
3. Subjects with active perianal fistula and non active luminal CD defined by a CDAI ≤ 200.
4. Subjects with perianal fistula confirmed by clinical assessment and MRI.
5. Subjects aged between 18 and 70, both male and female.
6. All subjects and their partners were not planning to have a child from screening to the end of the trial and agreed to use effective non-drug contraception during the trial.
7. Subjects failed to respond to adequate treatment with any of the conventional antibiotics, immunomodulatory drugs (including steroids), anti-tumor necrosis factor-α (TNF-α) monoclonal antibodies and other biological agents.

Exclusion Criteria:

1. Subjects with active infection evaluated by the investigator.
2. Subjects with Crohn's disease requiring immediate therapy.
3. Subjects with abscess or collections >2 cm.
4. Subjects with rectal and/or anal stenosis and/or active proctitis.
5. Subjects who treated with systemic steroids in the 4 weeks prior to stem cells administration.
6. Subjects with abnormal laboratory results: liver function: total bilirubin >=1.5 × ULN, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >=2 × ULN; renal function: creatinine clearance below 60 mL/minute calculated using Cockcroft-Gault formula or by serum creatinine >=1.5 × upper limit of normal (ULN).
7. Subjects with malignant tumors or a history of malignant tumors.
8. Subjects with severe, progressive, uncontrolled hepatic, hematological, gastrointestinal (except Crohn's disease), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral diseases.
9. Serum virology test (HBeAg, HCV antibody, HIV antibody, Treponema pallidum antibody) positive.
10. Subjects allergic to gentamicin sulfate, anesthetics or contrast media.
11. Subjects allergic to MRI contrast.
12. Subjects who has received stem cells in a previous clinical study or as a therapeutic agent.
13. Subjects who has major surgery or severe trauma within 6 months prior to the screening period.
14. Subjects who has received any investigational drug within 3 months prior to the screening.
15. Subjects deemed inappropriate by the investigator to participate in this clinical trial.
16. The female participant who is pregnant, or is lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Severity and incidence of adverse events | 28 days
  Severity and incidence of adverse events within 28 days after adiministration
Dose-limiting toxicity (DLT) | 84 days
  Exploration of dose-limiting toxicity (DLT)
Maximum tolerated dose (MTD) | 84 days
  Exploration of maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Perianal fistula healing | 84 days
  Change from baseline in Van Assche Score by MRI test. The score range was from 0 to 25. Higher score means more severe disease.
Crohn's Disease Activity Index (CDAI) score | 84 days
  Change from baseline in the Crohn's Disease Activity Index (CDAI) score. Higher score means more severe disease and especially severe disease was defined as a value of greater than 450.
Perianal Disease Activity Index (PDAI) | 84 days
  Change from baseline in Perianal Disease Activity Index (PDAI). Total score ranges from 0 to 20. Higher score means more severe disease.
Inflammatory Bowel Disease Questionnaire（IBDQ）score | 84 days
  Change from baseline in IBDQ score. Total score ranges from 32 to 224. Higher score means better quality of life.
VAS score | 84 days
  Change from baseline in pain score (VAS score).Total score ranges from 0 to 10. Higher score means more pain.
Anal sphincter function：Wexner incontinence score | 84 days
  Change from baseline in anal sphincter function, Wexner incontinence score,Total score ranges from 0 to 20. Higher score means more severe disease.
Anal sphincter function： rectal pressure | 84 days
  Change from baseline in rectal pressure，In healthy people, the pressure ranges from 60 to 150mmHg, with the internal sphincter pressure accounts for about 80% and external sphincter pressure accounts for 20%.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No